CLINICAL TRIAL: NCT00663702
Title: A Phase 3B Multi-center Open-Label Study to Evaluate the Safety of Abatacept in Subjects Who Switch From Intravenous to Subcutaneous Abatacept Therapy
Brief Title: Phase IIIB Switching From Intravenous to Subcutaneous Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IM101-185
Record Dates: First submitted 2008-04-18; First posted 2008-04-22 (Estimated); Results first posted 2012-03-26 (Estimated); Last update posted 2015-03-09 (Estimated); Status verified 2015-02

CONDITIONS: Arthritis, Rheumatoid
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Abatacept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Abatacept

INTERVENTIONS:
Drug: Abatacept — Subcutaneous injection, 125 mg/mL, once weekly, 48 months
  Other Names: Orencia; BMS-188667

SUMMARY:
The purpose of this study is to determine whether switching to subcutaneous administration of abatacept will be safe in participants with rheumatoid arthritis who previously received long-term therapy with intravenous abatacept

ELIGIBILITY:
Inclusion Criteria:

* Recruitment from 2 Bristol-Myers Squibb (BMS) studies (BMS IM101-029 [NCT00048581] and BMS IM101-102 [NCT00048568]).
* Completion of final quarterly dosing visit in NCT00048581 or NCT00048568 as follows: US and Canadian participants: Day 1821 visit; Taiwanese participants: Day 1905 visit; Mexican participants: Day 1989 visit.
* Agreement to participate in BMS IM101-185 (NCT00663702) on final quarterly dosing visit in NCT00048581 or NCT00048568 study as follows: US and Canadian participants: Day 1821 visit; Taiwanese participants: Day 1905 visit; Mexican participants: Day 1989 visit.
* At the time of completion of the NCT00048581 or NCT00048568 protocol, participant did not meet any criteria requiring their discontinuation.
* Drug stabilization requirements: Participants who received concomitant medications (disease-modifying antirheumatic drugs, corticosteroids, and nonsteroidal anti-inflammatory drugs) at the time of their last quarterly dosing visit for NCT00048581 or NCT00048568 were required to maintain stable dose levels from the time they signed consent until the end of the first 3 months (Day 85) of the current study.
* Willingness to self-inject study medication (abatacept) or allow a caregiver to inject study medication.
* Willingness to adhere to study visit schedule and comply with other protocol requirements.
* Male or female (not nursing or pregnant)genders, at least 18 years of age. Women of childbearing potential (WOCBP) must have been practicing adequate contraceptive measures during the study and for up to 10 weeks after the last infusion of study medication in such a manner that the risk of pregnancy was minimized. WOCBP must have had a negative serum or urine pregnancy test result (minimum sensitivity of 25 IU/L or equivalent units of human chorionic gonadotropin [HCG]) within 48 hours prior to the start of study medication.

Exclusion Criteria:

* The following treatment or therapies should not be started on or after the final quarterly dosing visit from the NCT00048581 or NCT00048568 study: Any biologic; immunoabsorption columns (such as Prosorba columns); mycophenolate mofetil; cyclosporin A or other calcineurin inhibitors; D-penicillamine; any live vaccines within 3 months of Day 1 or scheduled to receive a live vaccine during the course of the study
* Current symptoms of severe, progressive, or uncontrolled renal, hepatic, hematologic, gastrointestinal, pulmonary, cardiac, neurologic, or cerebral disease, or a concomitant medical condition that, in the opinion of the Investigator, might have placed the participation at unacceptable risk for study participation
* Any clinical laboratory test result that was considered to be abnormal or not within acceptable limits on the final quarterly dosing visit of NCT00048581 or NCT00048568. Screening laboratory test results for NCT00663702 were based on the Day 1821 visit of NCT00048581 or NCT00048568 for participants enrolled at sites in the US or Canada and on the Day 1989 visit of NCT00048568 for participants enrolled at sites in Mexico.
* Imprisonment or involuntarily incarceration for treatment of either a psychiatric or physical (eg, infectious disease) illness
* Impairment, incapacitation, inability to complete study-related assessments, or illiteracy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2008-05; Primary Completion 2009-12 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (29):
- United States (18):
  - Rheumatology Associates Of N. Al, P.C., Huntsville, Alabama
  - Allergy & Rheumatology Medical Clinic, Inc., La Jolla, California
  - Valerius Medical Group &Research Ctr. Of Greater Long Beach, Long Beach, California
  - Desert Medical Advances, Palm Desert, California
  - Inland Rheumatology Clinical Trials Inc., Upland, California
  - Arthritis & Rheumatic Disease Specialties, Aventura, Florida
  - Diagnostic Rheumatology And Research,Pc, Indianapolis, Indiana
  - Graves Gilbert Clinic, Bowling Green, Kentucky
  - Physician Research Collaboration, Llc, Lincoln, Nebraska
  - Innovative Health Research, Las Vegas, Nevada
  - The Center For Rheumatology, Llp, Albany, New York
  - The Arthritis Clinic & Carolina Bone & Joint, Charlotte, North Carolina
  - Unifour Medical Research, Hickory, North Carolina
  - Cincinnati Rheumatic Disease Study Group, Cincinnati, Ohio
  - Portland Rheumatology Clinic, Lake Oswego, Oregon
  - Rheumatic Disease Associates, Ltd., Willow Grove, Pennsylvania
  - Walter F. Chase, Md, Austin, Texas
  - Arthritis Centers Of Texas, Dallas, Texas
- Canada (6):
  - Local Institution, Edmonton, Alberta
  - Local Institution, St. John's, Newfoundland and Labrador
  - Local Institution, Kitchener, Ontario
  - Local Institution, Toronto, Ontario
  - Local Institution, Montreal, Quebec
  - Local Institution, Québec, Quebec
- Mexico (5):
  - Local Institution, Tijuana, Estado de Baja California
  - Local Institution, Guadalajara, Jalisco
  - Local Institution, Mexico City, Mexico City
  - Local Institution, Nuevo León, Nuevo León
  - Local Institution, San Luis Potosí City, San Luis Potosí

REFERENCES:
- [Derived] Alten R, Bingham CO 3rd, Cohen SB, Curtis JR, Kelly S, Wong D, Genovese MC. Antibody response to pneumococcal and influenza vaccination in patients with rheumatoid arthritis receiving abatacept. BMC Musculoskelet Disord. 2016 May 26;17:231. doi: 10.1186/s12891-016-1082-z. PMID 27229685

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 3 locations and 32 sites worldwide: United States (20 sites), Canada (6 sites), and Mexico (6 sites).
Pre-assignment Details: A total of 126 participants were enrolled, and 3 discontinued prior to study start due to failure to continue to meet study eligibility criteria.
Groups:
- Subcutaneous Abatacept, 125 mg (Prior Anti-TNF Failure): Participants with active rheumatoid arthritis, who previously received intravenous abatacept and failed therapy with antitumor necrosis factor (anti-TNF) in an earlier study (NCT00048581, or Bristol-Myers Squibb [BMS] IM101-029), received subcutaneous abatacept, 125 mg, once weekly for 3 months (to Day 85). Participants received the first dose of subcutaneous abatacept within 4 weeks of the last quarterly dosing visit of the preceding intravenous abatacept study.
- Subcutaneous Abatacept, 125 mg (Prior Methotrexate Failure): Participants with active rheumatoid arthritis, who previously received intravenous abatacept and showed an inadequate response to treatment with methotrexate in an earlier study (NCT00048568,or BMS IM101-102), received subcutaneous abatacept, 125 mg, once weekly for 3 months (to Day 85). Participants received the first dose of subcutaneous abatacept within 4 weeks of the last quarterly dosing visit of the preceding intravenous abatacept study.
Period: Overall Study
Arm/Group | Subcutaneous Abatacept, 125 mg (Prior Anti-TNF Failure) | Subcutaneous Abatacept, 125 mg (Prior Methotrexate Failure)
Started | 52 | 71
Completed | 34 | 61
Not Completed | 18 | 10
Not completed — Adverse Event | 8 | 4
Not completed — Withdrawal by Subject | 3 | 1
Not completed — Pregnancy | 0 | 1
Not completed — Lost to Follow-up | 3 | 0
Not completed — Death | 1 | 1
Not completed — Lack of Efficacy | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Subcutaneous Abatacept, 125 mg (Prior Anti-TNF Failure): Participants with active rheumatoid arthritis, who previously received intravenous abatacept and failed therapy with antitumor necrosis factor (anti-TNF) in an earlier study (NCT00048581, or BMS IM101-029), received subcutaneous abatacept, 125 mg, once weekly for 3 months (to Day 85). Participants received the first dose of subcutaneous abatacept within 4 weeks of the last quarterly dosing visit of the preceding intravenous abatacept study.
- Total: Total of all reporting groups
Arm/Group | Subcutaneous Abatacept, 125 mg (Prior Anti-TNF Failure) | Subcutaneous Abatacept, 125 mg (Prior Methotrexate Failure) | Total
Number analyzed (Participants) | 52 | 71 | 123
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.5 (10.2) | 52.8 (13.8) | 54.3 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 59 | 101
  Male | 10 | 12 | 22
Race/Ethnicity, Customized [Number; unit: Partcipants]
  White | 47 | 70 | 117
  Black/African American | 3 | 0 | 3
  American Indian/Alaska Native | 1 | 0 | 1
  Asian | 0 | 1 | 1
  Other | 1 | 0 | 1
Region of Enrollment [Number; unit: Participants]
  North America | 52 | 16 | 68
  South America | 0 | 55 | 55
Mean Baseline High Sensitivity C-Reactive Protein Level [Mean (Standard Deviation); unit: μg/mL] | 0.94 (0.65) | 0.92 (0.88) | 0.93 (0.79)
Mean Baseline 28 Joint Disease Activity Score (DAS 28) [Mean (Standard Deviation); unit: Score on a scale] — The DAS 28 is a 28-item joint disease activity score used to quantify disease expression and progression in rheumatoid arthritis. Severity is indicated with increasing item score on the scale with 0=no joints affected and 28=all joints affected.
  Score on a scale | 3.55 (1.20) | 3.28 (1.29) | 3.39 (1.26)
Mean Number of Tender Joints at Baseline [Mean (Standard Deviation); unit: Joints] | 9.1 (12.8) | 8.8 (12.4) | 8.9 (12.5)
Mean Number of Swollen Joints at Baseline [Mean (Standard Deviation); unit: Joints] | 5.4 (6.4) | 4.3 (5.9) | 4.8 (6.1)
Participant Weight at Baseline [Number; unit: Participants]
  Less than 60 kilograms | 9 | 14 | 23
  60-100 kilograms | 30 | 54 | 84
  Greater than 100 kilograms | 10 | 3 | 13
  Missing | 3 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Death as Outcome, Serious Adverse Events (SAEs), Treatment-related SAEs, SAEs Leading to Discontinuation, Treatment-related Adverse Events (AEs), AEs Leading to Discontinuation, and AEs of Interest (AEIs) at Day 85
Description: An AE is a new or worsening illness, sign, or symptom or a clinically significant abnormal laboratory test result occurring during the study, regardless of causality, and noted by the investigators. Systemic injection reaction occurring ≤ 24 hours after dosing.
Time Frame: Day 1 (Baseline) through Day 85
Population: All participants who received at least 1 dose of study medication
Measure: Number; unit: Participants
Groups:
- Subcutaneous Abatacept, 125 mg: Participants with active rheumatoid arthritis, who previously received intravenous abatacept and failed therapy with antitumor necrosis factor or showed an inadequate response to treatment with methotrexate in an earlier study, received subcutaneous abatacept, 125 mg, once weekly. Participants received the first dose of subcutaneous abatacept within 4 weeks of the last quarterly dosing visit of the preceding intravenous abatacept study.
Arm/Group | Subcutaneous Abatacept, 125 mg
Number analyzed (Participants) | 123
Participants
  Deaths | 0
  SAEs | 1
  Treatment-related SAEs | 0
  SAEs leading to discontinuation | 0
  Treatment-related AEs | 11
  AEs leading to discontinuation | 1
  AEIs: Infections | 20
  AEIs: Malignancy | 0
  AEIs: Automimmune disorders (prespecified) | 0
  AEIs: Injection reactions (prespecified) Local | 2
  AEIs: Injection reactions (prespecified) Systemic | 2

2. Secondary Outcome: Mean Trough Serum Concentration (Cmin) of Abatacept
Description: Cmin of abatacept was determined from serum samples.
Time Frame: Days 29, 85, 57, and 85
Population: All participants who received at least 1 dose of study medication. n=patients who had at least 1 pharmacokinetic sample drawn postbaseline
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | Subcutaneous Abatacept, 125 mg
Number analyzed (Participants) | 123
μg/mL
  Day 29 (n=116) | 34.31 (46)
  Day 57 (n=117) | 34.25 (48)
  Day 85 (n=118) | 33.78 (48)

3. Primary Outcome: Number of Participants With Death As Outcome, Serious Adverse Events (SAEs), Treatment-related SAEs, SAEs Leading to Discontinuation, Treatment-related Adverse Events (AEs), and AEs Leading to Discontinuation
Description: An AE is a new or worsening illness, sign, or symptom or a clinically significant abnormal laboratory test result occurring during the study, regardless of causality, and noted by the investigators.
Time Frame: Day 1 (Baseline) through 56 days past last day of subcutaneous injection in the cumulative study period
Population: All participants who received at least 1 dose of study medication
Measure: Number; unit: Participants
Arm/Group | Subcutaneous Abatacept, 125 mg
Number analyzed (Participants) | 123
Participants
  Deaths | 4
  SAEs | 43
  Treatment-related SAEs | 11
  SAEs leading to discontinuation | 8
  Treatment-related AEs | 60
  AEs leading to discontinuation | 11

4. Primary Outcome: Number of Participants With Hematology Laboratory Values Meeting the Criteria for Marked Abnormality
Description: LLN=lower limit of normal; ULN=upper limit of normal; preRx=pretreatment. Marked abnormality criteria: Hemoglobin (g/dL) >3 decrease from preRx. Hematocrit (%)<0.75*preRx. Erythrocytes (*10^6 c/uL) <0.75*preRx. Platelet count (*10^9 c/L) <0.67*LLN or 1.5*ULN or, if preRx<LLN, use <0.5*preRx and <100,000 mm^3. Leukocytes (*10^3 c/uL) <0.75*LLN or >1.25*ULN or, if preRx<LLN, use <0.8*preRx or >ULN or, if preRx>ULN, use >1.2*preRx or <LLN. Eosinophils >0.750*10^3 c/uL. Lymphocytes <0.750*10^3 c/uL or >7.50*10^3 c/uL.
Time Frame: Day 1 (Baseline) through 56 days past last day of subcutaneous injection in the cumulative study period
Population: All participants who received at least 1 dose of study medication. n=patients evaluable
Measure: Number; unit: Participants
Arm/Group | Subcutaneous Abatacept, 125 mg
Number analyzed (Participants) | 123
Participants
  Hemoglobin, low (n=120) | 7
  Hematocrit, low (n=119) | 4
  Erythrocytes, low (n=120) | 4
  Platelet count, low (n=120) | 2
  Leukocytes, low (n=120) | 2
  Leukocytes, high (n=120) | 3
  Eosinophils (absolute), high (n=122) | 12
  Lymphocytes (absolute), low (n=122) | 15

5. Primary Outcome: Number of Participants With Liver and Kidney Function Laboratory Values Meeting the Criteria for Marked Abnormality
Description: LLN=lower limit of normal; ULN=upper limit of normal; preRx=pretreatment. Marked abnormality criteria: Alkaline phosphatase (U/L) >2*ULN or if preRx>ULN, use 3*preRx. Alanine aminotransferase (U/L)>3*ULN or if preRx>ULN, use >4*preRx. G-glutamyl transferase (U/L)>2*ULN or if preRx>ULN, use >3*preRx. Blood urea nitrogen (mg/dL)>2*preRx. Creatinine (mg/dL)>1.5*preRx.
Time Frame: Day 1 (Baseline) through 56 days past last day of subcutaneous injection in the cumulative study period
Population: All participants who received at least 1 dose of study medication. n=patients evaluable
Measure: Number; unit: Participants
Arm/Group | Subcutaneous Abatacept, 125 mg
Number analyzed (Participants) | 123
Participants
  Alkaline phosphatase, high (n=120) | 1
  Aspartate aminotransferase, high (n=120) | 3
  Alanine aminotransferase, high (n=120) | 6
  G-glutamyl transferase, high (n=120) | 7
  Blood urea nitrogen, high (n=120) | 5
  Creatinine, high (n=120) | 11

6. Primary Outcome: Number of Participants With Electrolyte Laboratory Values Meeting the Criteria for Marked Abnormality
Description: LLN=lower limit of normal; ULN=upper limit of normal; preRx=pretreatment. Sodium: <0.95*LLN or >1.05*ULN or if preRx<LLN, <0.95*preRx or >ULN, or if preRx>ULN,>1.05*preRx or <LLN. Potassium,serum: <0.9*LLN or >1.1*ULN or if preRx<LLN, use <0.9*preRx or >ULN or if preRx>ULN, 1.1*preRx or <LLN. Phosphorus: 0.75*LLN or 1.25*ULN or, if preRx<LLN, <0.67*preRx or >ULN or, if preRx>ULN, <LLN.
Time Frame: Day 1 (Baseline) through 56 days past last day of subcutaneous injection in the cumulative study period
Population: All participants who received at least 1 dose of study medication. n=patients evaluable
Measure: Number; unit: Participants
Arm/Group | Subcutaneous Abatacept, 125 mg
Number analyzed (Participants) | 123
Participants
  Sodium, serum, low (mEq/L) (n=120) | 2
  Potassium, serum, low (mEq/L) (n=120) | 6
  Phosphorus, inorganic, low (mg/dL) (n=120) | 2

7. Primary Outcome: Number of Participants With Chemistry Laboratory Values Meeting the Criteria for Marked Abnormality
Description: LLN=lower limit of normal; ULN=upper limit of normal; preRX=pretreatment. Criteria for marked abnormality: .
Time Frame: Day 1 (Baseline) to up to 56 days past the last day of subcutaneous injection in the cumulative study period
Population: All participants who received at least 1 dose of study medication. n=patients evaluable
Measure: Number; unit: Participants
Arm/Group | Subcutaneous Abatacept, 125 mg
Number analyzed (Participants) | 123
Participants
  Glucose, serum, low (n=122) | 17
  Glucose, serum, high (n=122) | 12
  Glucose, serum, fasting, low (n=59) | 5
  Glucose, serum, fasting, high (n=59) | 3
  Protein, total, low (n=120) | 1
  Protein, total, high (n=120) | 1
  Albumin, low (n=120) | 3

8. Secondary Outcome: Percentage of Participants With A Positive Anti-abatacept Response (Based on Enzyme-linked Immunosorbent Assay [ELISA]) at Day 85
Description: Using the ELISA, any positive (titer of 400 or greater) postbaseline sample was classified as positive immunogenicity. The percentage of participants with at least 1 positive antibody response (anti-abatacept and/or anti-CTLA4-T) during the 85 days was tabulated by antibody specificity and overall.
Time Frame: Day 1 (Baseline) through Day 85
Population: All participants who received at least 1 subcutaneous abatacept injection and who had at least 1 immunogenicity result reported (on the corresponding assay) on subcutaneous abatacept treatment. n=patients evaluable
Measure: Number; unit: Percentage of participants
Arm/Group | Subcutaneous Abatacept, 125 mg
Number analyzed (Participants) | 122
Percentage of participants
  Anti-abatacept (n=85) | 8.2
  Anti-CTLA4-T9 (n=122) | 0.8

9. Secondary Outcome: Percentage of Participants With A Positive Anti-abatacept Response (Based on Electrochemiluminescence [ECL] Immunoassay) at Day 85
Description: Number of participants was tabulated using ECL assay with at least 1 positive abatacept-induced immunogenic response (CTLA4 and possibly Ig, Ig and/or Junction Region) in the first 85 days. Positive response (titers >10) included:
  * A missing baseline immunogenicity measurement and a positive immunogenicity response postbaseline
  * A negative baseline immunogenicity response and a positive immunogenicity response postbaseline
  * A positive baseline immunogenicity response and a positive immunogenicity response postbaseline that has a titer value strictly greater than the baseline titer value
Time Frame: Day 1 (Baseline) through Day 85
Population: as for outcome 8
Measure: Number; unit: Percentage of participants
Arm/Group | Subcutaneous Abatacept, 125 mg
Number analyzed (Participants) | 122
Percentage of participants | 0

10. Secondary Outcome: Mean Disease Activity Score 28 Based on C-reactive Protein (DAS 28-CRP) Scores Over Time
Description: The DAS 28-CRP is a measure of disease activity in rheumatoid arthritis (RA) and assesses the 28 joints RA commonly affects; the score includes the number of tender and swollen joints (out of 28), C-reactive protein level (a measure of inflammation in the blood), and the patient's global assessment of health (ranging from very good to very bad). DAS-CRP scores range from 0 to 10, with higher values indicating greater disease activity. Individual measures are fed into a complex mathematical formula to produce the overall DAS (a score greater than 5.1 implies active disease; less than 3.2, well controlled disease; and less than 2.6, remission.)
Time Frame: Day 1 (Baseline) through Day 1093
Population: All participants who received at least 1 dose of study medication
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- Subcutaneous Abatacept, 125 mg (Prior Anti-TNF Failure): Participants with active rheumatoid arthritis, who previously received intravenous abatacept and failed therapy with antitumor necrosis factor (anti-TNF) in an earlier study (NCT00048581, or Bristol-Myers Squibb [BMS] IM101-029), received subcutaneous abatacept, 125 mg, once weekly. Participants received the first dose of subcutaneous abatacept within 4 weeks of the last quarterly dosing visit of the preceding intravenous abatacept study.
- Subcutaneous Abatacept, 125 mg (Prior Methotrexate Failure): Participants with active rheumatoid arthritis, who previously received intravenous abatacept and showed an inadequate response to treatment with methotrexate in an earlier study (NCT00048568,or BMS IM101-102), received subcutaneous abatacept, 125 mg, once weekly. Participants received the first dose of subcutaneous abatacept within 4 weeks of the last quarterly dosing visit of the preceding intravenous abatacept study.
Arm/Group | Subcutaneous Abatacept, 125 mg (Prior Anti-TNF Failure) | Subcutaneous Abatacept, 125 mg (Prior Methotrexate Failure)
Number analyzed (Participants) | 52 | 71
Units on a scale
  Day 29 (n=50, 69) | 3.60 (1.24) | 2.95 (1.31)
  Day 57 (n=49, 69) | 3.36 (1.11) | 2.96 (1.37)
  Day 85 (n=49, 70) | 3.44 (1.14) | 2.91 (1.30)
  Day 169 (n=48, 71) | 3.45 (1.10) | 2.93 (1.29)
  Day 253 (n=46, 71) | 3.60 (1.33) | 3.01 (1.21)
  Day 365 (n=45, 70) | 3.51 (1.32) | 3.09 (1.25)
  Day 449 (n=43, 69) | 3.58 (1.33) | 3.21 (1.35)
  Day 533 (n=43, 68) | 3.51 (1.23) | 3.08 (1.43)
  Day 617 (n=41, 67) | 3.31 (1.20) | 3.16 (1.37)
  Day 729 (n=41, 67) | 3.30 (1.12) | 3.15 (1.26)
  Day 813 (n=39, 65) | 3.38 (1.17) | 2.81 (1.05)
  Day 897 (n=38, 65) | 3.41 (1.46) | 3.02 (1.19)
  Day 981 (n=38, 65) | 3.32 (1.37) | 3.02 (1.28)
  Day 1093 (n=34, 65) | 3.21 (1.26) | 3.10 (1.37)

11. Secondary Outcome: Percentage of Participants With Low Disease Activity Score (LDAS) and Disease Activity Score 28 Based on C-reactive Protein (DAS 28-CRP) Remission Over Time:
Description: LDAS is defined as DAS 28-CRP ≤3.2. DAS 28-CRP remission is defined as DAS 28-CRP <2.6. The DAS 28-CRP is a measure of disease activity in rheumatoid arthritis (RA) and assesses the 28 joints RA commonly affects; the score includes the number of tender and swollen joints (out of 28), C-reactive protein level (a measure of inflammation in the blood), and the patient's global assessment of health (ranging from very good to very bad). DAS-CRP scores range from 0 to 10, with higher values indicating greater disease activity. Individual measures are fed into a complex mathematical formula to produce the overall DAS (a score greater than 5.1 implies active disease; less than 3.2, well controlled disease; and less than 2.6, remission.)
Time Frame: Day 1 (Baseline) through Day 1093
Population: All participants who received at least 1 dose of study medication
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Subcutaneous Abatacept, 125 mg (Prior Anti-TNF Failure) | Subcutaneous Abatacept, 125 mg (Prior Methotrexate Failure)
Number analyzed (Participants) | 52 | 71
Percentage of participants
  LDAS Day 29 (n=50, 69) | 40.0 [26.4 to 53.6] | 68.1 [57.1 to 79.1]
  Remission Day 29 (n=50, 69) | 24.0 [12.2 to 35.8] | 50.7 [38.9 to 62.5]
  LDAS Day 57 (n=49, 69) | 44.9 [31.0 to 58.8] | 60.9 [49.4 to 72.4]
  Remission Day 57 (n=49, 69) | 26.5 [14.2 to 38.9] | 47.8 [36.0 to 59.6]
  LDAS Day 85 (n=49, 70) | 40.8 [27.1 to 54.6] | 64.3 [53.1 to 75.5]
  Remission Day 85 (n=49, 70) | 24.5 [12.4 to 36.5] | 48.6 [36.9 to 60.3]
  LDAS Day 169 (n=48, 71) | 39.6 [25.7 to 53.4] | 59.2 [47.7 to 70.6]
  Remission Day 169 (n=48, 71) | 25.0 [12.8 to 37.2] | 49.3 [37.7 to 60.9]
  LDAS Day 253 (n=46, 71) | 39.1 [25.0 to 53.2] | 66.2 [55.2 to 77.2]
  Remission Day 253 (n=46, 71) | 30.4 [17.1 to 43.7] | 42.3 [30.8 to 53.7]
  LDAS Day 365 (n=45, 70) | 40.0 [25.7 to 54.3] | 57.1 [45.5 to 68.7]
  Remission Day 365 (n=45, 70) | 33.3 [19.6 to 47.1] | 42.9 [31.3 to 54.5]
  LDAS Day 449 (n=43, 69) | 41.9 [27.1 to 56.6] | 53.6 [41.9 to 65.4]
  Remission Day 449 (n=43, 69) | 30.2 [16.5 to 44.0] | 43.5 [31.8 to 55.2]
  LDAS Day 533 (n=43, 68) | 37.2 [22.8 to 51.7] | 60.3 [48.7 to 71.9]
  Remission Day 533 (n=43, 68) | 23.3 [10.6 to 35.9] | 48.5 [36.7 to 60.4]
  LDAS Day 617 (n=41, 67) | 46.3 [31.1 to 61.6] | 53.7 [41.8 to 65.7]
  Remission Day 617 (n=41, 67) | 29.3 [15.3 to 43.2] | 43.3 [31.4 to 55.1]
  LDAS Day 729 (n=41, 67) | 41.5 [26.4 to 56.5] | 59.7 [48.0 to 71.4]
  Remission Day 729 (n=41, 67) | 29.3 [15.3 to 43.2] | 34.3 [23.0 to 45.7]
  LDAS Day 813 (n=39, 65) | 43.6 [28.0 to 59.2] | 69.2 [58.0 to 80.5]
  Remission Day 813 (n=39, 65) | 25.6 [11.9 to 39.3] | 46.2 [34.0 to 58.3]
  LDAS Day 897 (n=38, 65) | 50.0 [34.1 to 65.9] | 60.0 [48.1 to 71.9]
  Remission Day 897 (n=38, 65) | 34.2 [19.1 to 49.3] | 43.1 [31.0 to 55.1]
  DLAS Day 981 (n=38, 65) | 50.0 [34.1 to 65.9] | 64.6 [53.0 to 76.2]
  Remission Day 981 (n=38, 65) | 42.1 [26.4 to 57.8] | 46.2 [34.0 to 58.3]
  LDAS Day 1093 (n=34, 65) | 52.9 [36.2 to 69.7] | 58.5 [46.5 to 70.4]
  Remission Day 1093 (n=34, 65) | 41.2 [24.6 to 57.7] | 50.8 [38.6 to 62.9]

12. Secondary Outcome: Mean Health Assessment Questionnaire-Disability Index (HAQ-DI) Scores Over Time
Description: The HAQ-DI assesses patients' functional ability by rating their abilities over the previous week. At least 2 questions are asked from each of 8 categories: dressing and grooming, hygiene, arising, reach, eating, grip, walking, and common daily activities. Patients rate difficulty performing specific tasks: 0=without difficulty, 1=with some difficulty, 2=with much difficulty, and 3=unable to do. The sum of the categories is divided by the number of categories answered, yielding a score from 0-3.
Time Frame: Day 1 (Baseline) to Day 1093
Population: All participants who received at least 1 dose of study medication
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Subcutaneous Abatacept, 125 mg (Prior Anti-TNF Failure) | Subcutaneous Abatacept, 125 mg (Prior Methotrexate Failure)
Number analyzed (Participants) | 52 | 71
Units on a scale
  Day 29 (n=51, 69) | 0.98 (0.70) | 0.80 (0.67)
  Day 57 (n=50, 71) | 0.92 (0.68) | 0.80 (0.67)
  Day 85 (n=49, 71) | 0.92 (0.67) | 0.82 (0.69)
  Day 169 (n=49, 71) | 0.97 (0.67) | 0.87 (0.74)
  Day 253 (n=48, 71) | 0.97 (0.69) | 0.87 (0.73)
  Day 365 (n=46, 70) | 0.96 (0.66) | 0.85 (0.69)
  Day 449 (n=43, 69) | 0.97 (0.75) | 0.89 (0.69)
  Day 533 (n=43, 68) | 1.07 (0.71) | 0.94 (0.71)
  Day 617 (n=42, 67) | 0.99 (0.74) | 0.87 (0.69)
  Day 729 (n=42, 67) | 0.98 (0.74) | 0.90 (0.71)
  Day 813 (n=40, 66) | 1.02 (0.74) | 0.88 (0.68)
  Day 897 (n=39, 65) | 1.06 (0.75) | 0.89 (0.73)
  Day 981 (n=39, 65) | 1.02 (0.76) | 0.91 (0.69)
  Day 1093 (n=34, 65) | 0.96 (0.74) | 0.92 (0.74)

13. Primary Outcome: Participants With Urinalysis Values Meeting the Criteria for Marked Abnormality
Description: preRX=pretreatment. For all values analyzed (protein, urine; glucose, urine; blood, urine: leukocyte esterase, urine; white blood cells, urine; red blood cells, urine): If missing preRx, use >=2 or, if value >= 4, or if preRx=0 or 0.5, use >=2 or, if preRx= 1, use >=3 or, if preRx=2 or 3, use >=4.
Time Frame: Day 1 (Baseline) through 56 days past last day of subcutaneous injection in the cumulative study period
Population: All participants who received at least 1 dose of study medication. n=patients evaluable
Measure: Number; unit: Participants
Arm/Group | Subcutaneous Abatacept, 125 mg
Number analyzed (Participants) | 123
Participants
  Protein, urine, high (n=122) | 12
  Glucose, urine, high (n=122) | 8
  Blood, urine, high (n=122) | 28
  Leukocyte esterase, urine, high (n=95) | 32
  White blood cells, urine, high (n=103) | 64
  Red blood cells, urine, high (n=91) | 33

14. Primary Outcome: Number of Participants With Adverse Events of Special Interest
Description: AEs of special interest are AEs that may be associated with the use of immunomodulatory drugs, such as infections, malignancies, autoimmune disorders, and injection reactions (defined as local injection site reactions and systemic injection reactions occurring within 24 hours of subcutaneous injection).
Time Frame: Day 1 (Baseline) to up to 56 days past the last day of subcutaneous injection in the cumulative study period
Population: All participants who received at least 1 dose of study medication.
Measure: Number; unit: Participants
Arm/Group | Subcutaneous Abatacept, 125 mg
Number analyzed (Participants) | 123
Participants
  Infections | 96
  Malignancies | 7
  Prespecified autoimmune disorders | 7
  Prespecified systemic injection reactions | 14

15. Primary Outcome: Mean Sitting Systolic and Diastolic Blood Pressure (BP)
Description: BP was measured after the patient had been seated quietly for at least 5 minutes and recorded during the screening visit, during every office visit prior to administration of subcutaneous injections, and at study discharge or 7 days after the last dose for patients who terminated early.
Time Frame: Before injection on Days 1, 29, 57, 85, 169, 253, 365, 449, 533, 617, 729, 813, 897, 981, 1093, 1177, 1261, 1345, 1457, 1541, 1625, 1709, and 1821
Population: All participants who received at least 1 dose of study medication. n=patients evaluable
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Subcutaneous Abatacept, 125 mg
Number analyzed (Participants) | 123
mm Hg
  Sitting Systolic BP Day 1 | 121.6 (16.15)
  Sitting Systolic BP Day 29 (n=120) | 123.6 (16.08)
  Sitting Systolic BP Day 57 (n=120) | 123.9 (16.95)
  Sitting Systolic BP Day 85 (n=120) | 124.3 (16.62)
  Sitting Systolic BP Day 169 (n=116) | 124.0 (15.09)
  Sitting Systolic BP Day 253 (n=114) | 122.3 (14.58)
  Sitting Systolic BP Day 365 (n=114) | 124.1 (15.0)
  Sitting Systolic BP Day 449 (n=111) | 123.9 (15.80)
  Sitting Systolic BP Day 533 (n=108) | 123.5 (15.08)
  Sitting Systolic BP Day 617 (n=109) | 124.4 (16.03)
  Sitting Systolic BP Day 729 (n=108) | 125.2 (16.09)
  Sitting Systolic BP Day 813 (n=105) | 125.6 (16.04)
  Sitting Systolic BP Day 897 (n=102) | 122.8 (13.15)
  Sitting Systolic BP Day 981 (n=101) | 123.5 (15.44)
  Sitting Systolic BP Day 1093 (n=98) | 122.9 (13.46)
  Sitting Systolic BP Day 1177 (n=84) | 124.4 (13.66)
  Sitting Systolic BP Day 1261 (n=73) | 123.0 (15.29)
  Sitting Systolic BP Day 1345 (n=64) | 120.6 (12.27)
  Sitting Systolic BP Day 1457 (n=64) | 124.5 (13.17)
  Sitting Systolic BP Day 1541 (n=64) | 121.0 (13.75)
  Sitting Systolic BP Day 1625 (n=64) | 123.4 (14.71)
  Sitting Systolic BP Day 1709 (n=48) | 122.7 (15.55)
  Sitting Systolic BP Day 1821 (n=3) | 123.7 (15.18)
  Sitting Diastolic BP Day 1 (n=123) | 73.9 (8.83)
  Sitting Diastolic BP Day 29 (n=120) | 75.6 (9.28)
  Sitting Diastolic BP Day 57 (n=120) | 74.3 (8.82)
  Sitting Diastolic BP Day 85 (n=120) | 74.9 (10.37)
  Sitting Diastolic BP Day 169 (n=116) | 74.3 (9.19)
  Sitting Diastolic BP Day 253 (n=114) | 73.9 (9.96)
  Sitting Diastolic BP Day 365 (n=114) | 74.0 (9.98)
  Sitting Diastolic BP Day 449 (n=111) | 74.4 (9.53)
  Sitting Diastolic BP Day 533 (n=108) | 74.8 (10.08)
  Sitting Diastolic BP Day 617 (n=109) | 74.9 (9.72)
  Sitting Diastolic BP Day 79 (n=108) | 75.5 (9.83)
  Sitting Diastolic BP Day 813 (n=105) | 75.8 (10.20)
  Sitting Diastolic BP Day 897 (n=102) | 75.0 (10.23)
  Sitting Diastolic BP Day 981 (n=101) | 75.2 (9.35)
  Sitting Diastolic BP Day 1093 (n=98) | 76.2 (10.78)
  Sitting Diastolic BP Day1177 (n=84) | 77.6 (9.04)
  Sitting Diastolic BP Day 1261 (n=73) | 76.3 (9.94)
  Sitting Diastolic BP Day 1345 (n=64) | 75.4 (8.21)
  Sitting Diastolic BP Day 1457 (n=64) | 76.8 (7.14)
  Sitting Diastolic BP Day 1541 (n=64) | 75.6 (9.53)
  Sitting Diastolic BP Day 1625 (n=64) | 75.6 (9.36)
  Sitting Diastolic BP Day 1709 (n=48) | 75.2 (9.74)
  Sitting Diastolic BP Day 1821 (n=3) | 69.3 (8.14)

16. Primary Outcome: Mean Heart Rate
Description: Heart rate was measured after the patient had been seated quietly for at least 5 minutes and recorded during the screening visit, during every office visit prior to administration of subcutaneous injections, and at study discharge or 7 days after the last dose for patients who terminated early.
Time Frame: as for outcome 15
Population: All participants who received at least 1 dose of study medication. n=patients evaluable
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Subcutaneous Abatacept, 125 mg
Number analyzed (Participants) | 123
Beats per minute
  Day 1 | 74.2 (9.56)
  Day 29 (n=120) | 74.9 (8.35)
  Day 57 (n=120) | 74.6 (8.63)
  Day 85 (n=120) | 74.5 (8.90)
  Day 169 (n=119) | 73.6 (9.05)
  Day 253 (n=115) | 73.9 (9.74)
  Day 365 (n=114) | 73.8 (9.37)
  Day 449 (n=111) | 73.5 (9.12)
  Day 533 (n=109) | 72.7 (8.41)
  Day 617 (n=109) | 73.6 (9.83)
  Day 729 (n=108) | 74.2 (9.71)
  Day 813 (n=105) | 72.8 (7.76)
  Day 897 (n=102) | 72.4 (10.05)
  Day 981 (n=101) | 73.0 (8.90)
  Day 1093 (n=98) | 71.9 (9.07)
  Day 1177 (n=84) | 72.6 (8.33)
  Day 1261 (n=73) | 72.3 (9.41)
  Day 1345 (n=64) | 72.6 (8.02)
  Day 1457 (n=64) | 72.1 (7.78)
  Day 1541 (n=64) | 72.7 (8.90)
  Day 1625 (n=64) | 72.5 (8.73)
  Day 1709 (n=48) | 74.0 (9.78)
  Day 1821 (n=3) | 74.0 (6.24)

17. Primary Outcome: Mean Temperature
Description: Temperature was measured after the patient had been seated quietly for at least 5 minutes and recorded during the screening visit, during every office visit prior to administration of subcutaneous injections, and at study discharge or 7 days after the last dose for patients who terminated early.
Time Frame: as for outcome 15
Population: All participants who received at least 1 dose of study medication. n=patients evaluable
Measure: Mean (Standard Deviation); unit: Degrees Celsius
Arm/Group | Subcutaneous Abatacept, 125 mg
Number analyzed (Participants) | 123
Degrees Celsius
  Day 1 | 36.4 (0.49)
  Day 29 (n=120) | 36.4 (0.43)
  Day 57 (n=120) | 36.3 (0.40)
  Day 85 (n=120) | 36.4 (0.43)
  Day 169 (n=119) | 36.4 (0.41)
  Day 253 (n=115) | 36.4 (0.38)
  Day 365 (n=114) | 36.3 (0.39)
  Day 449 (n=111) | 36.4 (0.46)
  Day 533 (n=109) | 36.4 (0.38)
  Day 617 (n=109) | 36.4 (0.41)
  Day 729 (n=108) | 36.3 (0.33)
  Day 813 (n=105) | 36.3 (0.48)
  Day 897 (n=102) | 36.4 (0.36)
  Day 981 (n=101) | 36.4 (0.44)
  Day 1093 (n=98) | 36.3 (0.43)
  Day 1177 (n=84) | 36.3 (0.39)
  Day 1261 (n=73) | 36.3 (0.41)
  Day 1345 (n=64) | 36.3 (0.33)
  Day 1457 (n=64) | 36.3 (0.39)
  Day 1541 (n=64) | 36.2 (0.36)
  Day 1625 (n=64) | 36.2 (0.43)
  Day 1709 (n=48) | 36.2 (0.37)
  Day 1821 (n=3) | 36.7 (0.21)

ADVERSE EVENTS:
Arm/Group | Subcutaneous Abatacept, 125 mg
Serious Adverse Events (participants affected / at risk) | 43/123
Other Adverse Events (participants affected / at risk) | 101/123
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Subcutaneous Abatacept, 125 mg (N=123)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Colonic fistula (Gastrointestinal disorders) | 1
Diverticulitis (Infections and infestations) | 1
Lung adenocarcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pericardial effusion (Cardiac disorders) | 1
Angina pectoris (Cardiac disorders) | 1
Aphasia (Nervous system disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 1
Cervical dysplasia (Reproductive system and breast disorders) | 1
Myocardial ischaemia (Cardiac disorders) | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 1
Renal colic (Renal and urinary disorders) | 1
Bronchitis (Infections and infestations) | 1
Colitis (Gastrointestinal disorders) | 1
Coronary artery disease (Cardiac disorders) | 1
Hiatus hernia (Gastrointestinal disorders) | 2
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1
Brain neoplasm benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Appendicitis (Infections and infestations) | 1
Chest pain (General disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dengue fever (Infections and infestations) | 1
Ovarian cyst (Reproductive system and breast disorders) | 1
Pneumonia (Infections and infestations) | 4
Soft tissue infection (Infections and infestations) | 1
Coronary artery occlusion (Cardiac disorders) | 1
Diverticular perforation (Gastrointestinal disorders) | 1
Gastric polyps (Gastrointestinal disorders) | 1
Hip fracture (Injury, poisoning and procedural complications) | 2
Intestinal perforation (Gastrointestinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Sarcoidosis (Immune system disorders) | 1
Urosepsis (Infections and infestations) | 1
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Angina unstable (Cardiac disorders) | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cholecystitis infective (Infections and infestations) | 1
Cholelithiasis (Hepatobiliary disorders) | 2
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Device failure (General disorders) | 1
Gallbladder adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Gastroenteritis (Infections and infestations) | 1
Bundle branch block left (Cardiac disorders) | 1
Foot deformity (Musculoskeletal and connective tissue disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 4
Pancreatitis acute (Gastrointestinal disorders) | 1
Pancytopenia (Blood and lymphatic system disorders) | 2
Radius fracture (Injury, poisoning and procedural complications) | 1
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Subcutaneous Abatacept, 125 mg (N=123)
Cataract (Eye disorders) | 7
Diarrhoea (Gastrointestinal disorders) | 7
Fall (Injury, poisoning and procedural complications) | 9
Hypertension (Vascular disorders) | 10
Bronchitis (Infections and infestations) | 14
Gastritis (Gastrointestinal disorders) | 7
Nasopharyngitis (Infections and infestations) | 34
Nausea (Gastrointestinal disorders) | 9
Oedema peripheral (General disorders) | 9
Depression (Psychiatric disorders) | 7
Pharyngitis (Infections and infestations) | 7
Back pain (Musculoskeletal and connective tissue disorders) | 13
Cough (Respiratory, thoracic and mediastinal disorders) | 17
Headache (Nervous system disorders) | 10
Influenza like illness (General disorders) | 8
Sinusitis (Infections and infestations) | 10
Urinary tract infection (Infections and infestations) | 24
Conjunctivitis (Infections and infestations) | 9
Dizziness (Nervous system disorders) | 10
Gastroenteritis (Infections and infestations) | 9
Anaemia (Blood and lymphatic system disorders) | 9
Upper respiratory tract infection (Infections and infestations) | 30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.